CLINICAL TRIAL: NCT00250796
Title: Trial of Thalidomide, a- Interferon +/- Octreotide in Patients With Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Ian Rabinowitz, MD; Principal Investigator, University of New Mexico - CRTC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1400C
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-12

CONDITIONS: Liver; Cancer
Keywords: Phase II; Hepatocellular carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular | interventions — Thalidomide; Interferon-alpha; Interferons; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Thalidomide+alpha interferon
  Interventions: Drug: Thalidomide, alpha interferon
- Arm 2 (Experimental): Thalidomide+interferon+Octreotide
  Interventions: Drug: Thalidomide, interferon, Octreotide

INTERVENTIONS:
Drug: Thalidomide, alpha interferon — If the patient SSR status is negative, patients will not be given subcutaneous injections of octreotide (Sandostatin LAR) but will receive the thalidomide and alfa interferon only.
  Arms: Arm 1
Drug: Thalidomide, interferon, Octreotide — If SSR status is positive or unknown, patients will receive oral doses of thalidomide starting at 200mg a day and increasing to 800mg at increments of 200 per week depending on tolerance. They will also receive injections three times a week of alpha interferon and monthly injections of octreotide (Sandostatin LAR) 30 mg into their buttocks muscle..
  Other Names: Sandostatin LAR
  Arms: Arm 2

SUMMARY:
Primary Aim Determine the response rate and time to progression of the combination of thalidomide, interferon, and octreotide in patients with unresectable hepatocellular carcinoma (cancer of the liver that can't be treated surgically).

Secondary Aims

1. Determine the toxicity of this combination in this population.
2. Determine the survival of this patient cohort treated with the combination.
3. Determine the percent of patients with hepatocellular carcinoma who have a positive octreotide scan.

DETAILED DESCRIPTION:
The purpose of this study is to determine the response rate and time to progression of the combination of thalidomide, alfa interferon, and octreotide (Sandostatin LAR) in patients with unresectable hepatocellular carcinoma. If patients are eligible for and agree to take part in the study, they will be assigned to one of two treatment arms depending on SSR status. If SSR status is positive or unknown, patients will receive oral doses of thalidomide starting at 200mg a day and increasing to 800mg at increments of 200 per week depending on tolerance. They will also receive injections three times a week of alpha interferon and monthly injections of octreotide (Sandostatin LAR) 30 mg into their buttocks muscle..

If the patient SSR status is negative, patients will not be given subcutaneous injections of octreotide (Sandostatin LAR) but will receive the thalidomide and alfa interferon only.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of hepatocellular or radiographic evidence of a hepatic lesion consistent with hepatoma and an alpha feto protein >500 ng/ ml
2. The tumor is unresectable
3. Performance status of < 2.0
4. > 18 years of age
5. Informed consent to be signed by patient
6. No previous treatment with thalidomide, alpha interferon, or octreotide
7. The patient may have received previous chemotherapy either systemically or via the intra hepatic artery.
8. The patient may have had previous surgery or regional therapy such as intra tumoral injection of alcohol, cryosurgery, or radiofrequency ablation.
9. The patient must have measurable disease.
10. If female, the patient must have a negative pregnancy test and agree not to fall pregnant during this therapy.
11. Bilirubin <3 X ULN, AST/ALT<3 X ULN, creat<2, ANC>1.5, Platelet>75K
12. Patients may not have symptomatic cholelithiasis.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-09; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Determine the response rate and time to progression of the combination of thalidomide, interferon, and octreotide in patients with unresectable hepatocellular carcinoma. | Disease progression and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico